CLINICAL TRIAL: NCT05124561
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase III Clinical Trial on the Efficacy, Safety, and Immunogenicity of Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) for Inhalation (Ad5-nCoV-IH) in Adults Aged 18 Years and Above Who Have Received One Dose of Intramuscular Ad5-nCoV
Brief Title: Study to Evaluate the inHaled Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) On the Protective-Efficacy in Adults (SeiHOPE)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial protocol was not approved by the regulatory authorities.
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-AD5NCOV-IH-Ⅲ
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Inhalation; Ad5; Efficacy; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19; Respiratory Aspiration; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 6500 participants, Ad5-nCoV-IH, single dose, nebulized inhalation
  Interventions: Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH)
- Placebo group (Placebo Comparator): 6500 participants, placebo, single dose, nebulized inhalation
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (adenovirus type 5 vector) for Inhalation (Ad5-nCoV-IH) — Nebulized inhalation through the mouth
  Arms: Experimental group
Biological: Placebo — Nebulized inhalation through the mouth
  Arms: Placebo group

SUMMARY:
This phase III clinical trial is an endpoint-driven randomized, double-blind, parallel-controlled, multicenter clinical trial, and around 13,000 subjects aged 18 years and above who have previously received 1 dose of intramuscular Ad5-nCoV will be recruited. Volunteers should have been vaccinated with intramuscular Ad5-nCoV > 56 days prior to enrollment. All subjects will receive 1 dose of investigational vaccine or placebo through nebulized inhalation. The ratio of subjects in the vaccine group and placebo group is 1:1 and the efficacy and safety of the investigational vaccine will be followed up for 52 weeks after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers aged 18 years and above who have received 1 dose of intramuscular Ad5-nCoV > 56 days at the enrollment.
* Volunteers who have provided informed consent and signed the informed consent form.
* Volunteers who are able and willing to comply with the requirements of the clinical study protocol, and can complete the entire follow-up period of this study.

Exclusion Criteria:

* Allergic to the active ingredient, any non-active ingredient, or substances used in the manufacturing process, or developed an allergy to similar vaccines in the past.
* History of severe anaphylactic reaction to vaccines (e.g., acute anaphylactic reactions, angioedema, dyspnea).
* History or family history of seizures, epilepsy, encephalopathy, or psychosis.
* Severe nasal or oral diseases, such as acute rhinitis (sinusitis), allergic rhinitis, oral ulcers, throat redness, and swelling.
* History of a definite diagnosis of COVID-19.
* Positive SARS-CoV-2 N antibody rapid screening kit (IgG and IgM) results.
* Received COVID-19 vaccine other than Ad5-nCoV.
* Axillary temperature > 37.0°C.
* Severe cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, or severe hypertension and cannot be controlled by drugs.
* Lung function abnormalities such as asthma, chronic obstructive pulmonary disease, and pulmonary fibrosis.
* Acute febrile illness, symptoms of upper respiratory tract infection, or infectious diseases.
* Severe chronic diseases, or diseases of the progressive stage that cannot be steadily controlled, such as diabetes or thyroid disorders.
* Asplenia or functional asplenia.
* Thrombocytopenia or other coagulation disorder.
* Received immunosuppressant or immunomodulatory therapy (continuous oral or intravenous infusion for more than 14 days), anti-allergic therapy, cytotoxic therapy within the past 6 months. Inhalational and local steroids are allowed.
* Received blood products within 4 months before receiving the investigational vaccine.
* Received other vaccines within the past 14 days or plan to receive other vaccines 14 days after scheduled immunization with the investigational vaccine.
* Volunteers under antituberculous treatment or with active tuberculosis.
* Received blood/plasma products or immunoglobulin 60 days before immunization with the investigational vaccine or planned to receive blood/plasma products or immunoglobulin during the entire study period.
* Females who are positive for the urine pregnancy test, pregnant, or breastfeeding, or females who plan to conceive within 3 months (urine pregnancy test will only be performed in female volunteers of childbearing age).
* Volunteers who are judged by the investigator with any contradiction to the study protocol or affected the signing of informed consent due to various medical, psychological,social, or other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 cases. | Day 14 to 12 months post vaccination
  The efficacy of Ad5-nCoV-IH in preventing virologically confirmed (PCR positive) COVID-19 disease.
Incidence of SAE | Within 12 months post vaccination
  Evaluate the incidence of severe adverse events (SAE)

SECONDARY OUTCOMES:
Incidence of COVID-19 cases | Day 28 to 12 months post vaccination
  The efficacy of Ad5-nCoV-IH in preventing virologically confirmed (PCR positive) COVID-19 disease.
Incidence of severe COVID-19 cases | Day 14 and Day 28 to 12 months post vaccination
  Evaluate the efficacy of Ad5-nCoV in preventing severe COVID-19 disease caused by SARS-CoV-2 infection.
Incidence of COVID-19 cases in different age groups | Day 14 and Day 28 to 12 months post vaccination
  The efficacy of Ad5-nCoV-IH in preventing virologically confirmed (PCR positive) COVID-19 disease in participants between 18-59 years, and participants aged 60 years and above.
Incidence of Adverse Reactions (ARs) | Within 30 minutes post vaccination
  Incidence of ARs within 30 minutes post vaccination in the safety cohort.
Incidence of Adverse Reactions (ARs) | Within 14 days post vaccination
  Incidence of ARs within 14 days post vaccination in the safety cohort.
Incidence of Adverse Events (AEs) | Within 28 days post vaccination
  Incidence of AEs within 28 days post vaccination in the safety cohort.
Immunogenicity of S-RBD IgG antibody (ELISA method) | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  Seroconversion rate of S-RBD IgG antibody post vaccination.
Immunogenicity of S-RBD IgG antibody (ELISA method) | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  GMT of S-RBD IgG antibody post vaccination.
Immunogenicity of S-RBD IgG antibody (ELISA method) | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  GMI of S-RBD IgG antibody post vaccination.
Immunogenicity of neutralizing antibodies | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  Seroconversion rate of neutralizing antibodies post vaccination.
Immunogenicity of neutralizing antibodies | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  GMT of neutralizing antibodies post vaccination.
Immunogenicity of neutralizing antibodies | Day 14, Day 28, Week 24, and Week 52 post-vaccination
  GMI of neutralizing antibodies post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No